CLINICAL TRIAL: NCT03352414
Title: The ILEUS Study: A Phase 2 Randomized Controlled Trial Investigating Alvimopan for Enhanced Gastrointestinal Recovery After Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Phase 2 RCT of Alvimopan vs. Placebo After CRS/HIPEC
Acronym: ILEUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: stopped by sponsor
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Joel Baumgartner, Assistant Professor of Surgery, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 171044
Record Dates: First submitted 2017-11-18; First posted 2017-11-24 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Ileus
Keywords: HIPEC; peritoneal carcinomatosis
MeSH Terms: conditions — Ileus; Peritoneal Neoplasms | interventions — alvimopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alvimopan (Experimental): alvimopan 12 mg PO twice daily, starting POD 1 for the earlier of 7 days or hospital discharge
  Interventions: Drug: Alvimopan
- Placebo (Placebo Comparator): Placebo pill PO twice daily, starting POD 1 for the earlier of 7 days or hospital discharge
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alvimopan — alvimopan pill
  Other Names: Entereg
  Arms: Alvimopan
Drug: Placebo — placebo pill
  Other Names: Placebi
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the ability of alvimopan to reduce the time to return of bowel function in patients undergoing cytoreductive surgery and hyperthermic intraperitoneal chemotherapy. Half of the participants will receive alvimopan or and half will receive placebo immediately before and for up to seven days after surgery.

DETAILED DESCRIPTION:
Cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) is a surgical procedure to treat cancer that has spread to the lining of the abdominal cavity (peritoneal metastases). It is associated with a prolonged time for return of bowel function after surgery.

Alvimopan is a drug used to speed up the time for return of bowel function after surgery. It works by blocking the opioid receptors in the gastrointestinal tract, which normally slow down bowel function in patients receiving postoperative opioid pain medication. It has not previously been tested in patients undergoing CRS/HIPEC.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent.
* Scheduled to undergo open (non-minimally invasive) CRS/HIPEC.
* Scheduled to receive postoperative pain management with intravenous opioids.
* Age > 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Women of child-bearing potential with negative pregnancy test prior to initiating study drug dosing.

Exclusion Criteria:

* Greater than 7 days of consecutive opioid use immediately prior to scheduled surgery.
* Child-Pugh Class C hepatic impairment.
* End-stage renal disease (GFR < 15 mL/min/1.73 m2 and/or on peritoneal dialysis or hemodialysis).
* Complete mechanical bowel obstruction.
* Contraindication or inability to tolerate oral medication postoperatively.
* Presence of gastrointestinal ostomy after CRS/HIPEC.
* Pancreatic or gastric anastomosis performed during CRS/HIPEC.
* History of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition as alvimopan at the treating investigators discretion.
* Severe or uncontrolled medical disorder that would, in the investigator's opinion, impair ability to receive study treatment (i.e. uncontrolled diabetes, chronic renal disease, chronic pulmonary disease or active, uncontrolled infection, psychiatric illness/social situations that would limit compliance with study requirements).
* History of myocardial infarction in the 12 months prior to scheduled surgery.
* Pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Baumgartner, MD, MAS, Principal Investigator — UCSD
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Study was terminated early

REFERENCES:
- [Derived] Baumgartner JM, Chen R, Messer K, Veerapong J, Kelly KJ, Ramamoorthy S, Lowy AM. Alvimopan for Enhanced Gastrointestinal Recovery after Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy: A Randomized Controlled Trial. J Am Coll Surg. 2022 Nov 1;235(5):693-701. doi: 10.1097/XCS.0000000000000305. Epub 2022 Oct 17. PMID 36102565

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 84 participants were enrolled and randomized (constitute the safety population). All participants must later meet surgical eligibility for final allocation and analysis (n=62).
Period: Overall Study
Arm/Group | Alvimopan | Placebo
Started (Is the Randomized population meeting preoperative eligibility criteria (also called the Safety Population)) | 42 | 42
Allocated (Eligible by operative criteria (received additional postoperative study drug)) | 30 | 32
Completed | 30 | 32
Not Completed | 12 | 10
Not completed — Ineligible by operative criteria | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Alvimopan: Alvimpan Arm
- Placebo: Placebo Arm
- Total: Total of all reporting groups
Arm/Group | Alvimopan | Placebo | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Median (Full Range); unit: years] | 53 [27 to 73] | 61 [28 to 79] | 57 [27 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 12 | 34
  Male | 8 | 20 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to Return of Upper and Lower GI Function
Description: The later of the time from surgery that the participant first tolerates solid food and the time that the participant first passes a bowel movement.
Time Frame: from surgery to discharge (generally no longer than two weeks)
Population: Study was terminated early, preliminary data
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Alvimopan | Placebo
Number analyzed (Participants) | 30 | 32
hours | 117 [102 to 158] | 152 [134 to 204]

2. Secondary Outcome: Prolonged Ileus
Description: The proportion of patients who do not pass flatus or bowel movement greater than 7 days from the time of surgery.
Time Frame: from surgery to discharge (generally no longer than two weeks)
Population: Study was terminated early, preliminary data
Measure: Count of Participants; unit: Participants
Arm/Group | Alvimopan | Placebo
Number analyzed (Participants) | 30 | 32
Participants | 3 | 12

3. Secondary Outcome: Time to Return of Bowel Function Components
Description: The time from surgery until:
  * The time to first flatus
  * The time to first bowel movement
  * The time to tolerance of solid food
Time Frame: from surgery to discharge (generally no longer than two weeks)
Population: Study was terminated early, preliminary data
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Alvimopan | Placebo
Number analyzed (Participants) | 30 | 32
hours
  Time to first flatus | 64 [51 to 93] | 79 [63 to 97]
  Time to first BM | 67 [62 to 89] | 89 [71 to 114]
  Time to tolerance of solid food | 117 [102 to 158] | 149 [134 to 188]

4. Secondary Outcome: Time to Discharge
Description: The time from surgery until discharge order written.
Time Frame: from surgery to discharge (generally no longer than two weeks)
Population: Study was terminated early, preliminary data
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Alvimopan | Placebo
Number analyzed (Participants) | 30 | 32
hours | 188 [147 to 212] | 190 [187 to 236]

5. Secondary Outcome: Serious Adverse Events
Description: The number and proportion of serious adverse events.
Time Frame: up to 30 days from surgery
Population: From Safety population (n=84) Study was terminated early, preliminary data
Measure: Count of Participants; unit: Participants
Arm/Group | Alvimopan | Placebo
Number analyzed (Participants) | 42 | 42
Participants | 7 | 5

6. Secondary Outcome: Subgroup Analyses
Description: All primary and secondary outcomes will be measured in the following subgroups:
  * 0 vs. 1 or greater bowel anastomoses
  * 0 vs. 1 or greater visceral resections
  * high vs. low amount of postoperative opioid use
  * epidural vs. no epidural
Time Frame: up to 30 days from surgery
Population: Study was terminated early, data was not collected.
Arm/Group | Alvimopan | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days from the the time of surgery
Description: CTCAE v 4.03 (grade 3 or higher considered serious adverse event) All participants in the safety population (n=84) were included in the adverse event analysis. Per the protocol, this includes all randomized patients who took at least one dose of the study medication, including screen failures (at the time of surgery) after randomization and subjects withdrawn from the study.
Arm/Group | Alvimopan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 7/42 | 5/42
Other Adverse Events (participants affected / at risk) | 35/42 | 37/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alvimopan (N=42) | Placebo (N=42)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Rectal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Gastric Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Thromboembolic Event (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Wound Dehiscence (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alvimopan (N=42) | Placebo (N=42)
Non-Serious Adverse Events (Surgical and medical procedures) | 35 (35) | 37 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT03352414/Prot_SAP_000.pdf